CLINICAL TRIAL: NCT06725264
Title: TYK2 Inhibition in Granuloma Annulare (GA) and Cutaneous Sarcoidosis (CS): an Opportunity for Pathogenesis Directed Therapy
Brief Title: Tyrosine Kinase 2 (TYK2) for GA and CS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was rescinded.
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000038598
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Sarcoidosis; Granuloma Annulare
MeSH Terms: conditions — Sarcoidosis; Granuloma Annulare | interventions — deucravacitinib

STUDY DESIGN:
Intervention Model Description: Male and female subjects at least 18 years of age with moderate to severe granuloma annulare or cutaneous sarcoidosis affecting at least 5%body surface area.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Granuloma Annulare (Experimental): Participants with GA will receive the TYK2 inhibitor deucravacitinib 6mg twice daily
  Interventions: Drug: Deucravacitinib
- Cutaneous Sarcoidosis (Experimental): Participants with CS will receive the TYK2 inhibitor deucravacitinib 6mg twice daily
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — 6 mg twice daily
  Other Names: Sotyktu

SUMMARY:
To investigate the role of an oral TYK2 inhibitor for the treatment of patients with moderate to severe sarcoidosis with cutaneous involvement (CSAMI score of 10 or greater) and GA (defined as a BSA involvement of at least 5%), which are difficult to treat.

DETAILED DESCRIPTION:
Primary Objective To determine if TYK2 specific inhibition is effective in treating sarcoidosis and granuloma annulare (GA), problematic granulomatous inflammatory diseases which are difficult to treat.

Secondary Objective To determine the effect of treatment of participants' quality of life and on biomarkers of disease activity which often involves internal organ changes in sarcoidosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients 18 years old or older
* Diagnosis of GA or cutaneous sarcoidosis with supportive skin biopsy
* BSA involvement of at least 5% (GA) or CSAMI numerical score of at least 10 (sarcoidosis)
* If patients are on systemic therapies or phototherapy for their GA, they must discontinue these therapies with a washout period of 4 weeks and must remain off them during the study
* If patients are on topical therapies for their GA, they must discontinue these therapies with a washout period of 2 weeks and must remain off them during the study
* If patients are taking other systemic therapies for their sarcoidosis, they must be taking a stable dose of the other medication(s) for at least 3 months with no plans to change the regimen in the next 6 months. With the exception of methotrexate or low dose prednisone (20 mg or less per day), use of concomitant immunosuppressants, e.g. infliximab, azathioprine, etc., will not be permitted.
* For sarcoidosis, washout of topical medications will be for 2 weeks.
* Washout for oral medications will not be possible in most cases. Patients will be allowed to continue concomitant prednisone (up to 20 mg daily) or weekly methotrexate (up to 15 mg daily).
* Females of childbearing potential must agree to use birth control during the study and there must be a negative pregnancy test documented prior to starting the medication.
* Patients must be willing to have skin biopsies, blood collection, and total body photography and to comply with clinic visits

Exclusion Criteria:

* Age <18 years old
* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin)
* Patients known to be HIV or hepatitis B or C positive, or have an active, serious infection herpes simplex, herpes zoster, and pneumonia. This would also include localized infections.
* Patients with positive tuberculin skin test or positive QuantiFERON® TB test
* Patients with significant hepatic impairment
* Patients with moderate renal impairment
* Patients with uncontrolled peptic ulcer disease
* Patients with a history of deep vein thrombosis and/or pulmonary embolism and/or clotting disorder
* Patients with any history of myocardial infarction or stroke.
* Patients taking concomitant immunosuppressive medications, with the exception of methotrexate and/or low-dose prednisone, including but not limited to mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or TNF-α inhibitors
* Women of childbearing potential who are unable or unwilling to use birth control while taking the medication
* Women who are pregnant or nursing
* Current smoker or history of any tobacco use
* Patients over 50 who have the presence of cardiovascular risk factor
* Screening labs outside the normal range for parameters associated with potential risk for treatment under investigation. Including but not limited to:

  i. Platelets <150,000/mm3, ii. Absolute neutrophil count <1,000/mm3, iii. Hemoglobin levels <8 g/dL, iv. Absolute lymphocyte count <500/mm3
* Patients who are taking clinically significant inhibitors of both CYP2C19 and CYP2C9, or strong CYP2C19 or CYP2C9 inducers, as well as P-gp substrate where small concentration changes may lead to serious or life-threatening toxicities.
* Patients who have received a live vaccine. Patients should wait a minimum of 2 weeks, if recently vaccinated, prior to initiating treatment and should not receive a live vaccine during treatment or 2 weeks post-treatment.
* Patients with any medical, psychiatric, or social condition that is likely to unfavorably affect the risk-benefit of continued study participation, interfere with study compliance or confound safety or efficacy assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent change in the BSA involvement of GA | Baseline and 6 months post-treatment
  The percent change in the BSA involvement of GA after 6 months of treatment for participants with moderate to severe GA affecting at least 5% body surface area (BSA).
Percent change in the Cutaneous Sarcoidosis Activity and Morphology Instrument (CSAMI) score | Baseline and 6 months post-treatment
  The percent change in the CSAMI after 6 months of treatment. CSAMI evaluates the severity of sarcoidosis lesions in sarcoidosis participants across different body areas with separate scales for "Activity" (assessing inflammation, induration, surface changes, and area of involvement) and "Damage" (assessing post-inflammatory changes like scarring and dyspigmentation), resulting in a total Activity score ranging from 0 to 165 and a total Damage score from 0 to 22; with, higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Changes in molecular signatures in skin before and after treatment | Baseline and 6 months post-treatment
  Changes in molecular signatures in skin at baseline vs. after 6 months of treatment. RNA-sequencing will be used to examine transcriptional profiles in this skin.
Changes in molecular signatures in blood before and after treatment | Baseline and 6 months post-treatment
  Changes in molecular signatures in blood at baseline vs. after 6 months of treatment. A high throughput proteomic assay will be used to examine molecular profiles in the blood.
Changes in Skindex-16 (Skin related quality of life index) | Baseline and 6 months post-treatment
  Changes in Skindex-16 (Skin related quality of life index) baseline vs. after 6 months of treatment. This is a 16 item validated skin related Quality of Life questionnaire which will be administered by the study team to assess how GA affects the participants quality of life. Scores range from 0-96, higher scores indicating more significant impact on quality of life.
Changes in Granuloma Annulare Severity and Morphology Instrument (GASMI) score | Baseline and 6 months post-treatment
  Changes in GASMI score baseline vs. after 6 months of treatment. The Granuloma Annulare Severity and Morphology Instrument is a clinical severity scoring tool for GA. The score is determined by the study team who will examine the participants skin to determine the severity of the GA in different anatomic areas. Scores range from 0-165 with higher score indicating a worse outcome.
Organ involvement on whole body PET | Baseline and 6 months post-treatment
  Percent change in organ involvement using whole body PET- CT imaging
King's Sarcoidosis Questionnaire (KSQ) | Baseline and 6 months post-treatment
  The KSQ is a self-administered questionnaire used to assess the health-related quality of life in patients with sarcoidosis. Total score range is from 0 to 100 with higher scores indicating better health status.
Sarcoidosis Fatigue Assessment Scale (FAS) | Baseline and 6 months post-treatment
  The FAS is a 10-item self-report questionnaire used to measure the severity of fatigue in individuals with sarcoidosis, where each item is rated on a 5-point Likert scale ranging from "never" to "always". Total score is calculated by summing up all responses with a total score range from 10 (minimal fatigue) to 50 (extreme fatigue). Higher scores indicate greater fatigue.
Rhinosinusitis Disability Index (RSDI) | Baseline and 6 months post-treatment
  The RSDI is a 30-item questionnaire used to assess the impact of rhinosinusitis on a patient's quality of life. Each question is rated on a scale from 0 ("never") to 4 ("always") with a total score ranging from 0 to 120. Higher scores indicate greater disability,

CONTACTS AND LOCATIONS:
Overall Officials: William Damsky, MD, Principal Investigator — Yale University
Locations (1):
- YCCI/Church Street Research Unit (CSRU), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No